CLINICAL TRIAL: NCT05402631
Title: Can Patient Expectations Influence Pain Reduction After Epidural Injections in Patients With Low Back Pain? An Observational Cohort Study
Brief Title: Can Patient Expectations Influence Pain Reduction After Epidural Injections in Patients With Low Back Pain?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Regionale di Lugano (Other)
Collaborators: Faculty of Biomedical Sciences, Università della Svizzera Italiana, Lugano, Switzerland (Unknown)
Responsible Party: Principal Investigator, Eva Koetsier MD PhD LLM, Principal Investigator, Ospedale Regionale di Lugano
Other Study IDs: The EXPECT study
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Expectations; Back Pain; Back Pain Lower Back Chronic; Satisfaction, Patient; Injections, Epidural; Injections, Periradicular; Pain, Back
Keywords: Expectations; Influence of Expectations on Outcome; Back Pain; Epidural Injections; Periradicular Injections
MeSH Terms: conditions — Back Pain; Patient Satisfaction | interventions — Injections, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New patient with lower back pain
  Interventions: Procedure: Epidural Injection; Procedure: Periradicular Injection
- known patient with lower back pain
  Interventions: Procedure: Epidural Injection; Procedure: Periradicular Injection

INTERVENTIONS:
Procedure: Epidural Injection — patient receives an epidural injection due to lower back pain
Procedure: Periradicular Injection — patient receives a periradicular injection due to lower back pain

SUMMARY:
Investigators hypothesize that patients with higher expectations regarding their epidural injection experience a higher pain reduction of their lower back pain and/or leg pain after an epidural injection. Patients' expectations of an epidural injection can influence their level of pain reduction. The primary objective of this study is to investigate the prognostic significance of patient expectations on pain reduction after epidural injections ('expected benefits', see under) in patients with low back pain and/or leg pain.

Investigators furthermore hypothesize that patients that have a higher match between their expectations of improvement and actual improvement are more satisfied. A secondary objective of this study is to investigate the prognostic significance of a high match between expectations of improvement and actual improvement on patient satisfaction of the treatment.

DETAILED DESCRIPTION:
Chronic low back pain (with or without lower extremity pain) is extremely common problem in primary care and the leading cause worldwide for disability. Approximately 70 to 85% of the western population will develop low back pain at least once during their lifetime.

Low back pain is pain, muscle tension, or stiffness localized below the costal margin and above the inferior gluteal folds, with or without sciatica, and is defined as chronic when it persists for 12 weeks or more. The burden on the economy of low back pain were estimated at €2.6 billion and the direct medical costs at 6.1% of the total healthcare expenditure in Switzerland. Multiple modalities of treatments are utilized in managing chronic low back pain including analgesics, physiotherapy, injections, acupuncture, or surgery. Intralaminar and transforaminal lumbar epidural injections of corticosteroids have shown to be effective in patients with chronic low back pain and or leg pain.

Several studies demonstrated how patients' expectations are important predictors of the postsurgical health outcome. Patients' expectations are frequently studied as prognostic factors in knee and hip arthroplasty. It was shown that patients undergoing elective orthopaedic surgery whose expectations were fulfilled were found to be more satisfied with the overall treatment as compared to those whose expectations were not fulfilled. Furthermore, it was found that there is a robust small positive association between patients' positive preoperative expectations and better patient-reported postoperative outcomes. Investigators hypothesize that patient expectations of the pain treatment is also an important predictor of the pain reduction after epidural injections in patients with low back pain and/or leg pain. Therefore, the aim of this study is to investigate the prognostic significance of patient expectations on pain reduction after epidural injections in patients with low back pain and/or leg pain.

ELIGIBILITY:
Inclusion criteria

Subjects fulfilling all of the following inclusion criteria are eligible for the investigation:

* Age > 18 years old.
* Patients treated with a fluoroscopic guided lumbar epidural injection (transforaminal/translaminar/caudal) for back and/or leg pain

Exclusion criteria The presence of any one of the following exclusion criteria will lead to the exclusion of the subject

* patients who did not complete the questionnaires
* patient did not sign the general consent form (EOC_M-AFRI-001/A)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of our pain management center that get a transforaminal, translaminar or caudal injection of the spine.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of the average pain severity | 10 days after injection
  The reduction of the average pain severity score of the Brief Pain Inventory Short form [Time Frame: 10 days after injection in comparison to baseline]. Brief Pain Inventory (BPI) Short form will be used to assess pain intensity after lumbar epidural injection. BPI assess for pain and its scale is measured between 0 - 10, where '0' indicates no pain and '10' indicates severe pain in the last 24 hours. A decrease in the BPI score of 2 or more from the baseline score is considered clinically significant and indicates an improvement in severity of the patient's pain.15 We will examine the prognostic significance of patient expectations ('expected benefits', see under) on pain reduction after epidural injections in patients with low back pain and/or leg pain.

SECONDARY OUTCOMES:
Brief Pain Inventory Short form: average pain interference score | 10 days after injection
  BPI average pain interference score assesses the interference the pain has on the patient's functioning. BPI interference is measured between 0-10, where '0' indicates no interference and '10' indicates severe interference with functioning
The reduction of the immediate pain severity score of the Brief Pain Inventory Short form | 1 hour after injection
  Again the scale is measured between 0 - 10, where '0' indicates no pain and '10' indicates severe pain. A decrease in the BPI score of 2 or more from the baseline score is considered clinically significant and indicates an improvement in severity of the patient's pain
Patient Global Impression of Change (PGIC) | 10 days after injection
  The PGIC rating is increasingly being used for determining clinically important change in measures such as ratings of pain. This scale is designed to quantify patient's improvement or deterioration over time, usually either to determine the effect of an intervention or to chart the clinical course of a condition. The scales ask that a person assess his or her current health status, recall that status at a previous time-point, and then calculate the difference between the two.
Patients' satisfaction | 10 days after injection
  o This scale is designed to quantify patient's satisfaction with the treatment. Patients will be asked to define the one number that best shows how satisfied they are with the results of their pain treatment. Its scale is measured between 0 - 10, where '0' indicates extremely dissatisfied and '10' indicates extremely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Koetsier, PhD, Study Director — Faculty of Biomedical Sciences, Università della Svizzera Italiana, Lugano, Switzerland; Valeria Scheiwiller, Principal Investigator — Faculty of Biomedical Sciences, Università della Svizzera Italiana, Lugano, Switzerland
Locations (1):
- Faculty of Biomedical Sciences, Università della Svizzera Italiana, Lugano, Switzerland, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Urits I, Burshtein A, Sharma M, Testa L, Gold PA, Orhurhu V, Viswanath O, Jones MR, Sidransky MA, Spektor B, Kaye AD. Low Back Pain, a Comprehensive Review: Pathophysiology, Diagnosis, and Treatment. Curr Pain Headache Rep. 2019 Mar 11;23(3):23. doi: 10.1007/s11916-019-0757-1. PMID 30854609
- [Result] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Result] Hurwitz EL, Randhawa K, Yu H, Cote P, Haldeman S. The Global Spine Care Initiative: a summary of the global burden of low back and neck pain studies. Eur Spine J. 2018 Sep;27(Suppl 6):796-801. doi: 10.1007/s00586-017-5432-9. Epub 2018 Feb 26. PMID 29480409
- [Result] Last AR, Hulbert K. Chronic low back pain: evaluation and management. Am Fam Physician. 2009 Jun 15;79(12):1067-74. PMID 19530637
- [Result] Andersson GB. Epidemiological features of chronic low-back pain. Lancet. 1999 Aug 14;354(9178):581-5. doi: 10.1016/S0140-6736(99)01312-4. PMID 10470716
- [Result] Chou R, Deyo R, Friedly J, Skelly A, Hashimoto R, Weimer M, Fu R, Dana T, Kraegel P, Griffin J, Grusing S, Brodt ED. Nonpharmacologic Therapies for Low Back Pain: A Systematic Review for an American College of Physicians Clinical Practice Guideline. Ann Intern Med. 2017 Apr 4;166(7):493-505. doi: 10.7326/M16-2459. Epub 2017 Feb 14. PMID 28192793
- [Result] Wieser S, Horisberger B, Schmidhauser S, Eisenring C, Brugger U, Ruckstuhl A, Dietrich J, Mannion AF, Elfering A, Tamcan O, Muller U. Cost of low back pain in Switzerland in 2005. Eur J Health Econ. 2011 Oct;12(5):455-67. doi: 10.1007/s10198-010-0258-y. Epub 2010 Jun 5. PMID 20526649
- [Result] Bredow J, Bloess K, Oppermann J, Boese CK, Lohrer L, Eysel P. [Conservative treatment of nonspecific, chronic low back pain : Evidence of the efficacy - a systematic literature review]. Orthopade. 2016 Jul;45(7):573-8. doi: 10.1007/s00132-016-3248-7. German. PMID 27075679
- [Result] Abdi S, Datta S, Trescot AM, Schultz DM, Adlaka R, Atluri SL, Smith HS, Manchikanti L. Epidural steroids in the management of chronic spinal pain: a systematic review. Pain Physician. 2007 Jan;10(1):185-212. PMID 17256030
- [Result] Falco FJ, Irwin L, Zhu J. Lumbar spine injection and interventional procedures in the management of low back pain. Clin Occup Environ Med. 2006;5(3):655-702, vii-viii. doi: 10.1016/j.coem.2006.04.001. PMID 16963381
- [Result] Brunner M, Schwarz T, Zeman F, Konig M, Grifka J, Benditz A. Efficiency and predictive parameters of outcome of a multimodal pain management concept with spinal injections in patients with low back pain: a retrospective study of 445 patients. Arch Orthop Trauma Surg. 2018 Jul;138(7):901-909. doi: 10.1007/s00402-018-2916-y. Epub 2018 Mar 7. PMID 29511801
- [Result] Auer CJ, Glombiewski JA, Doering BK, Winkler A, Laferton JA, Broadbent E, Rief W. Patients' Expectations Predict Surgery Outcomes: A Meta-Analysis. Int J Behav Med. 2016 Feb;23(1):49-62. doi: 10.1007/s12529-015-9500-4. PMID 26223485
- [Result] Ng Kuet Leong VS, Kastner A, Petzke F, Przemeck M, Erlenwein J. The influence of pain expectation on pain experience after orthopedic surgery: an observational cohort study. Minerva Anestesiol. 2020 Oct;86(10):1019-1030. doi: 10.23736/S0375-9393.20.14084-7. Epub 2020 Jul 1. PMID 32613811
- [Result] Laferton JAC, Oeltjen L, Neubauer K, Ebert DD, Munder T. The effects of patients' expectations on surgery outcome in total hip and knee arthroplasty: a prognostic factor meta-analysis. Health Psychol Rev. 2022 Mar;16(1):50-66. doi: 10.1080/17437199.2020.1854051. Epub 2020 Dec 21. PMID 33228474
- [Result] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521